CLINICAL TRIAL: NCT02763826
Title: Optimizing Current and Electrode Montage for Transcranial Direct Current Stimulation in Stroke Patients
Acronym: COBRE_JIpro3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00022248
Record Dates: First submitted 2015-01-23; First posted 2016-05-05 (Estimated); Results first posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Stroke
Keywords: Transcranial Direct Current Stimulation; tDCS
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Determine the Optimal tDCS current (Experimental): We will invesitigate the optimal curent in range of 1 mA to 4 mA. We hypothesize that 4 mA is tolerable, safe and can induce the highest level of cortical excitability in the lesional motor cortex.
  Interventions: Device: transcranial direct current stimulation
- Determine the optimal tDCS electrode montage (Experimental): We hypothesize that the bi-hemispheric stimulation with anodal stimulation on the lesional hemisphere and simultaneous cathodal stimulation on the non-lesional hemisphere induces more cortical excitability in the lesional hemisphere than either anodal stimulation on the affected hemisphere or cathodal stimulation on non-lesional hemisphere alone.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — brain stimulation using progressively increasing amounts of direct currents and in a variety of electrode montages
  Other Names: tdcs

SUMMARY:
The purpose of this study is to determine the optimal transcranial direct current stimulation (tDCS) amplitude and electrode montage that is both safe and efficacious

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that can modulate cortical excitability of targeted brain regions. Various studies have investigated tDCS use in stroke patients with motor impairments (cumulatively about 200 cases). Although these studies are mostly "proof of concept" with small sample size, they do suggest that tDCS may improve motor function. However these two questions have not been addressed systematically:

1. What is the optimal current for stroke patients?
2. What is the optimal tDCS electrode montage for stimulation?

This proposal lays the scientific foundation for systematic application of tDCS in stroke recovery research by progressively increasing tDCS currents and montages that are both safe and efficacious in population with stroke.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old with a first-ever ischemic stroke that occurred at least 6 months ago;
* Finished rehabilitation therapy(including inpatient or outpatient Physical Therapy (PT) / Occupational Therapy (OT) / Speech Therapy (SP)) at least one month ago;
* Unilateral limb weakness with Fugl Meyer-Upper Extremity Scale score less than 56 (out of 66);
* Motor Evoked Potentials (MEP) is inducible on abductor pollicis brevis (APB) muscle on the affected side by TMS.

Exclusion Criteria:

* Primary intracerebral hematoma, or subarachnoid hemorrhage,
* Bihemispheric ischemic strokes;
* History of prior stroke or old infarct demonstrated on the CT or MRI or documented in medical records;
* Other concomitant neurological disorders affecting upper extremity motor function;
* Documented history of dementia before or after stroke;
* Documented history of uncontrolled depression or psychiatric disorder either before or after stroke which could affect their ability to participate in the experiment;
* Uncontrolled hypertension despite treatment, specifically Systolic blood pressure (SBP)/ Diastolic Blood Pressure (DBP) >= 180/100 mmHg at baseline;
* Presence of any MRI/tDCS/TMS risk factors: a) an electrically, magnetically or mechanically activated metal or nonmetal implant including cardiac pacemaker, intracerebral vascular clips or any other electrically sensitive support system; b) non-fixed metal in any part of the body, including a previous metallic injury to eye; c) pregnancy, since the effect of tDCS on the fetus is unknown; d) history of seizure disorder or post-stroke seizure; e) preexisting scalp lesion, bone defect or hemicraniectomy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wuwei Feng, MD, MS, Principal Investigator — MEDICAL UNIVERSITY OF SOUTH CAROL
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chhatbar PY, Chen R, Deardorff R, Dellenbach B, Kautz SA, George MS, Feng W. Safety and tolerability of transcranial direct current stimulation to stroke patients - A phase I current escalation study. Brain Stimul. 2017 May-Jun;10(3):553-559. doi: 10.1016/j.brs.2017.02.007. Epub 2017 Feb 27. PMID 28279641

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part 1 was a 3+3 dose-escalation study, which allowed up to 6 participants at a given dose escalation step. Part 2 was a montage effect study, which was a cross-over study requiring 18 participants to finish the study (by completing 3 visits). Participants enrolled in Part 1 were allowed to be enrolled in Part 2, but repeat participation in the same part by the same subject was not allowed.
Groups:
- 1 mA Bihemispheric tDCS: Subjects will get tDCS at a current of 1 mA with bihemispheric montage
- 2 mA Bihemispheric tDCS: Subjects will get tDCS at a current of 2 mA with bihemispheric montage
- 2.5 mA Bihemispheric tDCS: Subjects will get tDCS at a current of 2.5 mA with bihemispheric montage
- 3 mA Bihemispheric tDCS: Subjects will get tDCS at a current of 3 mA with bihemispheric montage
- 3.5 mA Bihemispheric tDCS: Subjects will get tDCS at a current of 3.5 mA with bihemispheric montage
- 4 mA Bihemispheric tDCS: Subjects will get tDCS at a current of 4 mA with bihemispheric montage
- 4 mA Anodal tDCS: Subjects will get tDCS at a current of 4 mA with anodal montage
- 4 mA Cathodal tDCS: Subjects will get tDCS at a current of 4 mA with cathodal montage
Period: Part 1 Dose Escalation, 1 mA
Arm/Group | 1 mA Bihemispheric tDCS | 2 mA Bihemispheric tDCS | 2.5 mA Bihemispheric tDCS | 3 mA Bihemispheric tDCS | 3.5 mA Bihemispheric tDCS | 4 mA Bihemispheric tDCS | 4 mA Anodal tDCS | 4 mA Cathodal tDCS
Started | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 Dose Escalation, 2 mA
Arm/Group | 1 mA Bihemispheric tDCS | 2 mA Bihemispheric tDCS | 2.5 mA Bihemispheric tDCS | 3 mA Bihemispheric tDCS | 3.5 mA Bihemispheric tDCS | 4 mA Bihemispheric tDCS | 4 mA Anodal tDCS | 4 mA Cathodal tDCS
Started | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 Dose Escalation, 2.5 mA
Arm/Group | 1 mA Bihemispheric tDCS | 2 mA Bihemispheric tDCS | 2.5 mA Bihemispheric tDCS | 3 mA Bihemispheric tDCS | 3.5 mA Bihemispheric tDCS | 4 mA Bihemispheric tDCS | 4 mA Anodal tDCS | 4 mA Cathodal tDCS
Started | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 Dose Escalation, 3 mA
Arm/Group | 1 mA Bihemispheric tDCS | 2 mA Bihemispheric tDCS | 2.5 mA Bihemispheric tDCS | 3 mA Bihemispheric tDCS | 3.5 mA Bihemispheric tDCS | 4 mA Bihemispheric tDCS | 4 mA Anodal tDCS | 4 mA Cathodal tDCS
Started | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 Dose Escalation, 3.5 mA
Arm/Group | 1 mA Bihemispheric tDCS | 2 mA Bihemispheric tDCS | 2.5 mA Bihemispheric tDCS | 3 mA Bihemispheric tDCS | 3.5 mA Bihemispheric tDCS | 4 mA Bihemispheric tDCS | 4 mA Anodal tDCS | 4 mA Cathodal tDCS
Started | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 Dose Escalation, 4 mA
Arm/Group | 1 mA Bihemispheric tDCS | 2 mA Bihemispheric tDCS | 2.5 mA Bihemispheric tDCS | 3 mA Bihemispheric tDCS | 3.5 mA Bihemispheric tDCS | 4 mA Bihemispheric tDCS | 4 mA Anodal tDCS | 4 mA Cathodal tDCS
Started | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 Montage Effect, 1st Intervention
Arm/Group | 1 mA Bihemispheric tDCS | 2 mA Bihemispheric tDCS | 2.5 mA Bihemispheric tDCS | 3 mA Bihemispheric tDCS | 3.5 mA Bihemispheric tDCS | 4 mA Bihemispheric tDCS | 4 mA Anodal tDCS | 4 mA Cathodal tDCS
Started | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 Montage Effect, 2nd Intervention
Arm/Group | 1 mA Bihemispheric tDCS | 2 mA Bihemispheric tDCS | 2.5 mA Bihemispheric tDCS | 3 mA Bihemispheric tDCS | 3.5 mA Bihemispheric tDCS | 4 mA Bihemispheric tDCS | 4 mA Anodal tDCS | 4 mA Cathodal tDCS
Started | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 Montage Effect, 3rd Intervention
Arm/Group | 1 mA Bihemispheric tDCS | 2 mA Bihemispheric tDCS | 2.5 mA Bihemispheric tDCS | 3 mA Bihemispheric tDCS | 3.5 mA Bihemispheric tDCS | 4 mA Bihemispheric tDCS | 4 mA Anodal tDCS | 4 mA Cathodal tDCS
Started | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 mA Bihemispheric tDCS: Participants received 1 mA Bihemispheric tDCS
- 2 mA Bihemispheric tDCS: Participants received 2 mA Bihemispheric tDCS
- 2.5 mA Bihemispheric tDCS: Participants received 2.5 mA Bihemispheric tDCS
- 3 mA Bihemispheric tDCS: Participants received 3 mA Bihemispheric tDCS
- 3.5 mA Bihemispheric tDCS: Participants received 3.5 mA Bihemispheric tDCS
- 4 mA Bihemispheric tDCS: Participants received 4 mA Bihemispheric tDCS
- Crossover - 4mA Bihemisphere tDCS and 4 mA Anodal tDCS and 4mA Cathodal tDCS: Stroke subjects will each receive one of three stimulation montages
- Total: Total of all reporting groups
Arm/Group | 1 mA Bihemispheric tDCS | 2 mA Bihemispheric tDCS | 2.5 mA Bihemispheric tDCS | 3 mA Bihemispheric tDCS | 3.5 mA Bihemispheric tDCS | 4 mA Bihemispheric tDCS | Crossover - 4mA Bihemisphere tDCS and 4 mA Anodal tDCS and 4mA Cathodal tDCS | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 13 | 31
Age, Categorical [Count of Participants; unit: Participants] — Population: Dose escalation does not include Crossover period, Crossover period foes not include Dose Escalation period.
  Participants
    Dose Escalation: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 18
    Dose Escalation: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Dose Escalation: Between 18 and 65 years | 2 | 3 | 3 | 2 | 3 | 3 | 0 | 16
    Dose Escalation: >=65 years | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
    Crossover: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 13
    Crossover: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Crossover: Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9
    Crossover: >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Dose escalation does not include Crossover period, Crossover period foes not include Dose Escalation period.
  Participants
    Dose Escalation: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 18
    Dose Escalation: Female | 1 | 0 | 2 | 2 | 1 | 1 | 0 | 7
    Dose Escalation: Male | 2 | 3 | 1 | 1 | 2 | 2 | 0 | 11
    Crossover: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 13
    Crossover: Female | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
    Crossover: Male | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Dose escalation does not include Crossover period, Crossover period foes not include Dose Escalation period.
  Participants
    Dose Escalation: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 18
    Dose Escalation: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Dose Escalation: Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Dose Escalation: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Dose Escalation: Black or African American | 0 | 1 | 1 | 2 | 2 | 1 | 0 | 7
    Dose Escalation: White | 2 | 2 | 2 | 1 | 1 | 2 | 0 | 10
    Dose Escalation: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Dose Escalation: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Crossover: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 13
    Crossover: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Crossover: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Crossover: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Crossover: Black or African American | 0 | 00 | 0 | 0 | 0 | 0 | 7 | 7
    Crossover: White | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
    Crossover: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Crossover: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Dose Escalation | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 18
  United States: Crossover Period | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Response
Description: Major response is any of the following:
  * Second degree scalp burn at the site of electrode pad; or
  * Seizure; or
  * New lesion(s) on Diffusion Weighted Imaging (DWI) sequence of MRI scan and the lesion(s) not explained by any other cause(s) or decreased Apparent Diffusion Coefficient (ADC) under the electrode stimulating motor cortex area;
  * Discontinuation of subject from the study due to any of above.
  In a 3+3 design, 3 subjects are recruited for a given tDCS dose level. The trial is stopped if ≥2 of 3 subjects at a given tDCS dose level show major response. If only 1 of 3 subjects shows major response, 3 more subjects are recruited at a given tDCS dose level and a major response in any of them will stop the trial. Otherwise, same procedure is followed for the next tDCS dose level. Maximum tolerable dose will be the tDCS dose at the level before stopping of the trial.
Time Frame: Immediately after intervention on the day of tDCS application
Measure: Count of Participants; unit: Participants
Arm/Group | 1 mA Bihemispheric tDCS | 2 mA Bihemispheric tDCS | 2.5 mA Bihemispheric tDCS | 3 mA Bihemispheric tDCS | 3.5 mA Bihemispheric tDCS | 4 mA Bihemispheric tDCS | 4 mA Anodal tDCS | 4 mA Cathodal tDCS
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 21 | 18 | 19
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 years, 4 months
Groups:
- 1 mA Bihemispheric tDCS: Subjects will receive tDCS at 1 mA with bihemispheric montage
- 2 mA Bihemispheric tDCS: Subjects will receive tDCS at 2 mA with bihemispheric montage
- 2.5 mA Bihemispheric tDCS: Subjects will receive tDCS at 2.5 mA with bihemispheric montage
- 3 mA Bihemispheric tDCS: Subjects will receive tDCS at 3.0 mA with bihemispheric montage
- 3.5 mA Bihemispheric tDCS: Subjects will receive tDCS at 3.5 mA with bihemispheric montage
- 4 mA Bihemispheric tDCS: Subjects will receive tDCS at 4 mA with bihemispheric montage
- 4 mA Anodal tDCS: Subjects will receive tDCS at 4 mA with anodal montage
- 4 mA Cathodal tDCS: Subjects will receive tDCS at 4 mA with cathodal montage
Arm/Group | 1 mA Bihemispheric tDCS | 2 mA Bihemispheric tDCS | 2.5 mA Bihemispheric tDCS | 3 mA Bihemispheric tDCS | 3.5 mA Bihemispheric tDCS | 4 mA Bihemispheric tDCS | 4 mA Anodal tDCS | 4 mA Cathodal tDCS
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 1/3 | 0/21 | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/21 | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/21 | 0/18 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT02763826/Prot_SAP_000.pdf